CLINICAL TRIAL: NCT01990521
Title: Screening Male BRCA Mutation Carriers: Effectiveness of Multispectral 3T Magnetic Resonance Imaging
Brief Title: Prostate Screening Study Using MRI in BRCA Carriers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Sunnybrook Regional Cancer Centre (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Women's College Hospital (Other)
Responsible Party: Principal Investigator, Danny Vesprini, MD, MSc, FRCPC, Radiation Oncologist, Toronto Sunnybrook Regional Cancer Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 500-2013
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MS3TMRI / TRUS Guided Biopsy (Experimental)
  Interventions: Procedure: MS3TMRI / TRUS Guided Biopsy; Device: MS3TMRI / TRUS Guided Biopsy

INTERVENTIONS:
Procedure: MS3TMRI / TRUS Guided Biopsy — Patients would undergo MS3TMRI and then have a transrectal ultrasound (TRUS) biopsy performed within one month after the MRI. The initial cores would be obtained using TRUS without MRI information (TRUSBx). During the same biopsy session, the MS3TMRI information would be given to the physician performing the biopsy and additional cores specifically targeted to suspicious areas would be performed (MS3TMRI-TRUSBx).
Device: MS3TMRI / TRUS Guided Biopsy — Multispectral 3T MRI (MS3TMRI) is a device that uses a 3T MRI system without an endorectal receiver coil and with a surface phased array coil. 3T MRI in addition to established computer aided diagnosis (CAD) has been used to perform guided biopsies in an active surveillance population and demonstrated a positive predictive value and negative predictive value of 83% and 81%.
  A recently completed a study looking at repeat prostate biopsies in men followed on an active surveillance population at Sunnybrook has shown that the PPV of MS3TMRI guided biopsy to be 85%, while the negative predictive value was 100% (Haider, Vesprini and Milot, unpublished).
  Other Names: Multispectral 3T MRI; Transrectal Ultrasound

SUMMARY:
Men with a BRCA1 or BRCA2 mutation are at increased risk for early onset, aggressive prostate cancer compared to men in the general population.

Standard of care screening for men with a BRCA mutation includes PSA testing and digital rectal examination (DRE), the same as with men in the general population.

This study is being done to assess whether there is value in using MRI as a screening tool to detect prostate cancer at an earlier stage than may otherwise be detected using standard of care screening (PSA, DRE). It is unclear whether MRI has utility as a screening tool in this specific population at high risk for aggressive disease.

DETAILED DESCRIPTION:
To determine the value of using Multispectral 3T MRI (MS3TMRI) for prostate cancer screening in men with a high risk of developing early onset aggressive prostate cancer given known BRCA1 or BRCA2 mutation carrier status, with no prior prostate cancer diagnosis, independent of baseline PSA levels.

* Determine the prevalence of prostate cancer in BRCA1 and BRCA2 mutation carriers independent of baseline PSA levels.
* To evaluate the accuracy of tumor targeting based on MRI and ultrasound (US) tumor co-localization. To evaluate the sensitivity, specificity, PPV, NPV, and accuracy of an automated computer aided diagnosis method (CAD) applied to MS3TMRI in the prediction of zonal biopsy results for the presence or absence of a significant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Male Hereditary Cancer Research Program at Sunnybrook Health Sciences Center.
* Have positive genetic testing for a pathogenic BRCA1 or BRCA2 mutation.
* Clinically eligible for and willing to undergo ultrasound biopsy within 4 weeks after the MRI.
* Be 50 years of age or older.

Exclusion Criteria:

* Claustrophobia
* Contraindication to MRI
* Contraindication to receiving low molecular weight MRI contrast agent
* Previously diagnosed with prostate cancer

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2025-09 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prostate MRI in BRCA carriers | 2 years (January 2016)
  Measure of prostate MRI to determine the PPV of MRI for detection of actionable prostate cancer

SECONDARY OUTCOMES:
Prostate cancer in BRCA carriers | 2 years January 2016
  Prevalence of any prostate cancer compared to actionable cancer in men with a BRCA1 or BRCA2 mutation independent of serum PSA value.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J Vesprini, MD, MSc, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada